CLINICAL TRIAL: NCT02757625
Title: Phase 3, Multi-center, Single-arm, Open-label Study Evaluating The Efficacy, Safety, And Pharmacokinetics Of Da-9501 (Dexmedetomidine Hydrochloride) In Pediatric Subjects In The Intensive Care Unit
Brief Title: Study of DA-9501 In Pediatric Subjects In The Intensive Care Unit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Maruishi Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0801017; ZIN-DEX-1506 (Other: Alias Study Number)
Record Dates: First submitted 2016-04-11; First posted 2016-05-02 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-05

CONDITIONS: ICU Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DA-9501 (Experimental): A single vial contains an injection solution with 2 mL of dexmedetomidine hydrochloride solution (100 µg/mL as dexmedetomidine) dissolved in physiological saline
  Interventions: Drug: Dexmedetomidine hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine hydrochloride — * 45 weeks CGA to < 6 years old: Maintenance infusion will be started at 0.2 µg/kg/h. The infusion rate will be adjusted within a range of 0.2 to 1.4 µg/kg/h according to the pediatric subject's sedative state
  * 6 years old to < 17 years old: Maintenance infusion will be started at 0.2 µg/kg/h. The infusion rate will be adjusted within a range of 0.2 to 1.0 µg/kg/h according to the pediatric subject's sedative state

SUMMARY:
To evaluate the efficacy, safety, and pharmacokinetics of dexmedetomidine given as continuous IV infusion in pediatric subjects [≥ 45 weeks CGA (corrected gestational age) to <17 years old] requiring sedation under intensive care unit

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose consent is obtained in writing prior to the clinical trial from a guardian after a full explanation. For subjects over 7 years old, it is desirable that an informed assent is also obtained from the pediatric subject him/herself when possible.
2. Subjects aged ≥45 weeks CGA to <17 years old at time of consent. No restriction on sex of subject.
3. [Elective surgical cases] Subjects classified as American Society of Anesthesiologists (ASA) (ASA physical status classification) Class I to III by preoperative diagnosis.
4. [Elective surgical cases] Subjects who require at least 6 hours of respiratory management with intubation under intensive care from immediately after surgery and are anticipated to require sedation.
5. [Medical ICU cases] Subjects who require at least 24 hours of respiratory management with intubation under intensive care and are anticipated to require sedation. For medical ICU cases, sedatives used prior to treatment with the investigational product should be discontinued before the start of treatment with the investigational product.
6. If a subject is a female of childbearing potential, she should not be pregnant or possibly pregnant, or lactating.

Exclusion Criteria:

1. Subjects who are judged by investigator or sub-investigator to have a neurological disease that will make sedation assessment difficult, such as:

   * Subjects with brain damage which is expected to increase intracranial pressure due to trauma or central nervous system disease
   * Subjects with cerebral palsy, autism, severe mental retardation, etc.
   * Subjects with paralysis due to continuous administration of a muscle relaxant or due to a spinal injury of class T5 or higher.
2. Subjects with 2nd or 3rd degree heart block during the tests at the screening visit (excluding subjects using a pacemaker).
3. Subjects with any of the following low blood pressure levels during the tests at the screening visit:

   * Age ≥ 45 weeks CGA to < 1 year old: Systolic Blood Pressure (SBP) <70 mmHg
   * Age ≥ 1 year old to < 10 years old: SBP < 70 + (2 x age in years) mmHg
   * Age ≥ 10 years old to < 17 years old: SBP < 90 mmHg
4. Subject of bradycardia (≤10th centile of heart rate for healthy children) during the physical examination at screening period.
5. Subjects with ALT ≥100 U/L during the laboratory tests at the screening visit.
6. Subjects in whom dexmedetomidine or other alfa 2 receptor agonists, alfa 2 receptor antagonists and drug that may be used in this study are contraindicated.
7. Subjects who may need a sedative or analgesic (including narcotics) other than dexmedetomidine, midazolam or fentanyl during treatment with the investigational product.
8. Subjects who have acute febrile illness [with a temperature (core or tympanic) ≥ 38.0°Centigrade] at the screening visit.
9. Subjects who received other investigational product within 30 days before baseline or subjects who will participate in other study that uses an investigational product during the study period.
10. Subjects who received dexmedetomidine within 48 hours before baseline.
11. Subjects who, in the opinion of the investigator or sub-investigator, may be at increased risk to the subject due to the conduct of the study or may have a disease or factor which will probably preclude the obtainment of sufficient study data.
12. Subjects for whom, in the opinion of the investigator or sub-investigator, risks involved with administration of dexmedetomidine outweigh its benefits (e.g., >2 doses of vasopressor due to cardiogenic shock).
13. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Sponsor's employees directly involved in the conduct of the study.

Ages: 45 Weeks to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Japan (12):
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Shikoku Medical Center for Children and Adults, Zentsujichó, Kagawa-ken
  - Osaka Women's and Children's Hospital, Izumi, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Shizuoka Children's Hospital, Shizuoka

REFERENCES:
- [Derived] Takeuchi M, Nemoto S, Suzuki Y, Takahashi N, Takenaka N, Takata A, Kobayashi M. Age-Specific Dose Regimens of Dexmedetomidine for Pediatric Patients in Intensive Care Following Elective Surgery: A Phase 3, Multicenter, Open-Label Clinical Trial in Japan. Pediatr Crit Care Med. 2021 Nov 1;22(11):e546-e557. doi: 10.1097/PCC.0000000000002730. PMID 33813550
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ZIN-DEX-1506&StudyName=Phase+3%2C+Multi-center%2C+Single-arm%2C+Open-label+Study+Evaluating+The+Efficacy%2C+Safety%2C+And+Pharmacokinetics+Of+Da-9501+%28dexmedetomidine+Hydrochloride%29+In+Pediatric+Subjects+In+The+Intensive+Care+Unit
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0801017&StudyName=Phase+3%2C+Multi-center%2C+Single-arm%2C+Open-label+Study+Evaluating+The+Efficacy%2C+Safety%2C+And+Pharmacokinetics+Of+Da-9501+%28dexmedetomidine+Hydrochloride%29+In+Pediatric+Subjects+In+The+Intensive+Care+Unit

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: >=45 Weeks CGA to <12 Months: Participants with age between >=45 weeks corrected gestation age (CGA) to <12 months received 0.2 microgram per kilogram per hour (mcg/kg/h) of dexmedetomidine infusion for up to 28 days. The infusion rate was adjusted from 0.2 to 1.4 mcg/kg/h as per pediatric participant's sedative state.
- Dexmedetomidine: >=12 Months to <24 Months: Participants with age between >=12 months to <24 months received 0.2 mcg/kg/h of dexmedetomidine infusion for up to 28 days. The infusion rate was adjusted from 0.2 to 1.4 mcg/kg/h as per pediatric participant's sedative state.
- Dexmedetomidine: >=2 Years to <6 Years: Participants with age between >=2 years to <6 years received 0.2 mcg/kg/h of dexmedetomidine infusion for up to 28 days. The infusion rate was adjusted from 0.2 to 1.4 mcg/kg/h as per pediatric participant's sedative state.
- Dexmedetomidine: >=6 Years to <17 Years: Participants with age between >=6 years to <17 years received 0.2 mcg/kg/h of dexmedetomidine infusion for up to 28 days. The infusion rate was adjusted from 0.2 to 1.4 mcg/kg/h as per pediatric participant's sedative state.
Period: Overall Study
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years
Started | 14 | 18 | 19 | 12
Completed | 14 | 18 | 17 | 12
Not Completed | 0 | 0 | 2 | 0
Not completed — Investigator's discretion | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who have received at least one dose of the study drug.
Groups:
- Dexmedetomidine: >=45 Weeks CGA to <12 Months: Participants with age between >=45 weeks CGA to <12 months received 0.2 microgram per mcg/kg/h of dexmedetomidine infusion for up to 28 days. The infusion rate was adjusted from 0.2 to 1.4 mcg/kg/h as per pediatric participant's sedative state.
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Total
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.1 (2.1) | 16.9 (3.6) | 45.7 (14.6) | 112.1 (37.9) | 41.3 (41.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 5 | 27
  Male | 6 | 11 | 12 | 7 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 18 | 19 | 12 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Did Not Require a Rescue Sedative Within 24 Hours of Dosing of Study Drug
Description: Percentage of participants who did not require rescue medication for Sedation (Midazolam) based on the data of investigator's judgement and State Behavioral Scale (SBS) (which was a sedation assessment instrument for intubated participants and its score ranges from 2 to -3, where 2= agitated, 1= restless and difficult to calm, 0= awake and able to calm, -1= responsive to gentle touch or voice, -2= responsive to noxious stimuli and -3= unresponsive. During intubation [placement of a flexible plastic tube into the trachea to maintain an open airway or to serve as a conduit through which to administer certain drugs], the target sedation depth by SBS was -2 to 0, where higher score indicated more responsive and after extubation [removal of endotracheal tube], the target sedation depth was -1 to 0, where higher score indicated more responsive) were reported.
Time Frame: From start of study drug administration on Day 1 up to 24 hours of study drug dosing or at the conclusion of mechanical ventilation or the end of study drug administration, whichever is earliest (up to maximum of 28 days)
Population: FAS included all participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dexmedetomidine: All Participants: Participants with age between >=45 weeks CGA to <17 years received 0.2 microgram per mcg/kg/h of dexmedetomidine infusion for up to 28 days. The infusion rate was adjusted from 0.2 to 1.4 mcg/kg/h as per pediatric participant's sedative state.
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
percentage of participants | 78.6 [51.7 to 93.2] | 66.7 [43.6 to 83.9] | 78.9 [56.1 to 92.0] | 91.7 [62.5 to 100.0] | 77.8 [66.0 to 86.4]

2. Secondary Outcome: Percentage of Participants Who Did Not Require Administration of a Rescue Analgesic Within 24 Hours of Dosing of Study Drug
Description: Percentage of participants who did not require administration of a rescue analgesic (Fentanyl) in addition to administration of the study drug based on investigator's judgement were reported.
Time Frame: as for outcome 1
Population: FAS included all participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
percentage of participants | 85.7 [58.8 to 97.2] | 100.0 [79.3 to 100.0] | 94.7 [73.5 to 100.0] | 66.7 [38.8 to 86.4] | 88.9 [78.5 to 94.8]

3. Secondary Outcome: Total Amount of Rescue Sedative Administered Within 24 Hours of Dosing of Study Drug
Description: Total amount of rescue sedative (midazolam) administered Within 24 Hours of dosing of study drug.
Time Frame: as for outcome 1
Population: Analysis was performed on only rescued participants (defined as all participants who received any amount of rescue medication in the specified evaluation period).
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 3 | 6 | 4 | 1 | 14
milligrams (mg) | 0.882 (0.8282) | 3.188 (1.6935) | 2.469 (1.3975) | 1.960 | 2.401 (1.5793)

4. Secondary Outcome: Body Weight Adjusted Total Amount (Per Kg) of Rescue Sedative Taken Within 24 Hours of Dosing of Study Drug
Description: Total amount of rescue sedative (midazolam) required within 24 hours of dosing of study drug. Dose was adjusted for body weight (mg divided by kg).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 3 | 6 | 4 | 1 | 14
mg/kg | 0.135 (0.1160) | 0.353 (0.2219) | 0.142 (0.0668) | 0.100 (0) | 0.228 (0.1866)

5. Secondary Outcome: Total Amount of Rescue Analgesic Taken Within 24 Hours of Dosing of Study Drug
Description: Total amount of rescue sedative (fentanyl) required Within 24 Hours of dosing of study drug.
Time Frame: as for outcome 1
Population: Analysis was performed on only rescued participants (defined as all participants who received any amount of rescue medication in the specified evaluation period). Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 0 | 1 | 4 | 7
micrograms | 91.70 (78.772) |  | 97.50 (0) | 81.74 (15.754) | 86.84 (34.676)

6. Secondary Outcome: Body Weight Adjusted Total Amount of Rescue Analgesic Taken Within 24 Hours of Dosing of Study Drug
Description: Total amount of rescue analgesic (fentanyl) within 24 Hours of dosing of study drug. Dose was adjusted for body weight (mcg divided by kg).
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 0 | 1 | 4 | 7
mcg/kg | 15.00 (9.899) |  | 5.00 (0) | 3.78 (1.311) | 7.16 (6.789)

7. Secondary Outcome: Duration of Maintenance of Target Sedation Level Within 24 Hours of Dosing of Study Drug
Description: Time duration for which the target sedation level was maintained during the specified evaluation period within participants was reported. Target sedation level was analyzed by target sedation scores by using the SBS. SBS was a sedation assessment instrument for intubated participants and its score ranges from 2 to -3, where 2= agitated, 1= restless and difficult to calm, 0= awake and able to calm, -1= responsive to gentle touch or voice, -2= responsive to noxious stimuli and -3= unresponsive. During intubation (placement of a flexible plastic tube into the trachea to maintain an open airway or to serve as a conduit through which to administer certain drugs), the target sedation depth by SBS was -2 to 0, where higher score indicated more responsive and after extubation (removal of endotracheal tube), the target sedation depth was -1 to 0, where higher score indicated more responsive.
Time Frame: as for outcome 1
Population: FAS included all participants who received at least one dose of the study drug. Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 13 | 17 | 19 | 11 | 60
hours | 7.95 (7.191) | 3.89 (2.859) | 3.52 (5.495) | 2.96 (2.017) | 4.50 (5.112)

8. Secondary Outcome: Percentage of Maintenance Duration of Target Sedation Level Within 24 Hours of Dosing of Study Drug
Description: Percentage of time duration for which the target sedation level was maintained during the specified evaluation period within participants was reported. Target sedation level was analyzed by target sedation scores by using the state behavioral scale (SBS). SBS is a sedation assessment instrument and it's score ranges from 2 to -3, where 2= agitated, 1= restless and difficult to calm, 0= awake and able to calm, -1= responsive to gentle touch or voice, -2= responsive to noxious stimuli and -3= non-responsive. During intubation the target sedation depth by SBS was -2 to 0, where higher score indicated more responsive and after extubation, the target sedation depth was -1 to 0, where higher score indicated more responsive.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 13 | 17 | 19 | 11 | 60
percentage of time | 54.08 (31.825) | 60.97 (28.104) | 50.54 (27.898) | 62.25 (34.836) | 56.54 (29.911)

9. Secondary Outcome: Percentage of Participants Who Did Not Use a Rescue Sedative After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: Percentage of participants whose period of dosing of the investigational product exceeded 24 hours and who did not received rescue medication for Sedation (Midazolam) based on the data of investigator's judgement and SBS (which was a sedation assessment instrument for intubated participants and its score ranges from 2 to -3, where 2= agitated, 1= restless and difficult to calm, 0= awake and able to calm, -1= responsive to gentle touch or voice, -2= responsive to noxious stimuli and -3= unresponsive. During intubation [placement of a flexible plastic tube into the trachea to maintain an open airway or to serve as a conduit through which to administer certain drugs], the target sedation depth by SBS was -2 to 0, where higher score indicated more responsive and after extubation [removal of endotracheal tube], the target sedation depth was -1 to 0, where higher score indicated more responsive) were reported.
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: Participants from FAS population whose period of dosing of investigational product exceeded 24 hours.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 3
percentage of participants | 100.0 [29.0 to 100.0] |  | 100.0 [16.7 to 100.0] |  | 100.0 [38.3 to 100.0]

10. Secondary Outcome: Percentage of Participants Who Did Not Require Dosing of a Rescue Analgesic After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: Percentage of participants whose period of dosing of the investigational product exceeded 24 hours and who did not received rescue analgesic (Fentanyl) based on the investigator's judgement were reported.
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: Participants from FAS population whose period of dosing of investigational product exceeded 24 hours.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 3
percentage of participants | 100.0 [29.0 to 100.0] |  | 100.0 [16.7 to 100.0] |  | 100.0 [38.3 to 100.0]

11. Secondary Outcome: Total Amount of Rescue Sedative Taken After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: Total amount of rescue sedative (midazolam) administered after 24 hours of dosing of study drug.
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: as for outcome 3
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Body Weight Adjusted Total Amount of Rescue Sedative Taken After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: Total amount of rescue sedative (midazolam) required after 24 hours of dosing of study drug. Dose was adjusted for body weight (mg divided by kg).
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: Analysis was performed on only rescued participants (defined as all participants who received any amount of rescue sedative in the specified evaluation period).
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Total Amount of Rescue Analgesic Taken After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: Total amount of rescue analgesic (Fentanyl) administered by the participants after 24 hours of dosing of study drug.
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: as for outcome 3
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Body Weight Adjusted Total Amount of Rescue Analgesic Taken After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: Total amount of rescue analgesic (fentanyl) after 24 hours of dosing of study drug. Dose was adjusted for body weight (mcg divided by kg).
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: as for outcome 3
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Duration of Maintenance of Target Sedation Level After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: Time duration for which the target sedation level was maintained during the specified evaluation period within participants was reported. Target sedation level was analyzed by target sedation scores by using the state behavioral scale (SBS). SBS is a sedation assessment instrument for intubated participants and its score ranges from 2 to -3, where 2= agitated, 1= restless and difficult to calm, 0= awake and able to calm, -1= responsive to gentle touch or voice, -2= responsive to noxious stimuli and -3= unresponsive. During intubation (placement of a flexible plastic tube into the trachea to maintain an open airway or to serve as a conduit through which to administer certain drugs), the target sedation depth by SBS was -2 to 0, where higher score indicated more stability and after extubation (removal of endotracheal tube), the target sedation depth was -1 to 0, where higher score indicated more stability.
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: Participants from FAS population whose period of dosing of investigational product exceeded 24 hours.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 3
hours | 0.81 (0.672) |  | 0.92 (0) |  | 0.84 (0.479)

16. Secondary Outcome: Percentage of Maintenance Duration of Target Sedation Level After 24 Hours of Dosing of Study Drug Till End of Mechanical Ventilation
Description: as for outcome 8
Time Frame: After 24 hours of study drug dosing till end of mechanical ventilation (up to 28 days)
Population: Participants from FAS population whose period of dosing of investigational product exceeded 24 hours.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 3
percentage of time | 75.00 (35.355) |  | 100.00 (0) |  | 83.33 (28.868)

17. Secondary Outcome: Duration of Maintenance of Target Sedation Level After Extubation
Description: Time duration for which the target sedation level was maintained during the specified evaluation period within participants was reported. Target sedation level was analyzed by target sedation scores by using the state behavioral scale (SBS). SBS is a sedation assessment instrument for intubated participants and its score ranges from 2 to -3, where 2= agitated, 1= restless and difficult to calm, 0= awake and able to calm, -1= responsive to gentle touch or voice, -2= responsive to noxious stimuli and -3= unresponsive. During intubation (placement of a flexible plastic tube into the trachea to maintain an open airway or to serve as a conduit through which to administer certain drugs), the target sedation depth by SBS was -2 to 0, where higher score indicated more responsive and after extubation (removal of endotracheal tube), the target sedation depth was -1 to 0, where higher score indicated more responsive.
Time Frame: From extubation till end of treatment (6 hours after start of study drug dosing up to 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 16 | 10 | 58
hours | 11.68 (11.589) | 7.73 (7.543) | 7.60 (4.355) | 6.73 (5.036) | 8.42 (7.679)

18. Secondary Outcome: Percentage of Maintenance Duration of Target Sedation Level After Extubation
Description: as for outcome 8
Time Frame: From extubation till end of treatment (6 hours after start of study drug dosing up to 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 16 | 10 | 58
Percentage of time | 69.99 (28.260) | 53.93 (28.613) | 54.45 (30.805) | 55.82 (41.195) | 58.19 (31.829)

19. Secondary Outcome: Total Amount of Rescue Sedative Taken After Extubation
Description: Total amount of rescue sedative (Midazolam) administered by the participants after extubation.
Time Frame: From extubation till end of treatment (6 hours after start of study drug dosing up to 28 days)
Population: Analysis was performed on only rescued participants (defined as all participants who received any amount of rescue sedative in the specified evaluation period). Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 5
mg | 0.537 (0.3741) | 0.719 (0.3379) | 5.994 |  | 1.701 (2.4148)

20. Secondary Outcome: Body Weight Adjusted Total Amount of Rescue Sedative Taken After Extubation
Description: Total amount of rescue sedative (midazolam) administered by the participants after extubation. Dose was adjusted for body weight (mg divided by kg).
Time Frame: From extubation till end of treatment (6 hours after start of study drug dosing up to 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 5
mg/kg | 0.109 (0.0976) | 0.072 (0.0304) | 0.370 |  | 0.146 (0.1364)

21. Secondary Outcome: Total Amount of Rescue Analgesic Taken After Extubation
Description: Total amount of rescue analgesic (fentanyl) administered by the participants after extubation.
Time Frame: From extubation till end of treatment (6 hours after start of study drug dosing up to 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
mcg |  |  | 42.90 |  | 42.90

22. Secondary Outcome: Body Weight Adjusted Total Amount of Rescue Analgesic Taken After Extubation
Description: Total amount of rescue analgesic (fentanyl) administered by the participants after extubation. Dose was adjusted for body weight (mcg divided by kg).
Time Frame: From extubation till end of treatment (6 hours after start of study drug dosing up to 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
mcg/kg |  |  | 3.00 |  | 3.00

23. Secondary Outcome: Median Time to Conclusion of Mechanical Ventilation
Description: Time to conclusion of mechanical ventilation was defined as time duration from start of study drug administration until the end of mechanical ventilation.
Time Frame: Baseline (start of study drug dosing) until end of mechanical ventilation (up to 28 days)
Population: FAS: all participants who received at least one dose of the investigational product.
Measure: Median (Full Range); unit: hours
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
hours | 9.5 [6.3 to 17.5] | 6.0 [4.6 to 6.3] | 4.1 [3.0 to 6.0] | 4.5 [3.8 to 6.0] | 6.0 [4.8 to 6.2]

24. Other Pre Specified Outcome: Number of Participants With Treatment- Emergent Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to up to 28 days after end of study drug dosing (up to 56 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both non-serious adverse events (AEs) and SAEs.
Time Frame: Baseline up to 28 days after end of study drug dosing (up to 56 days)
Population: Safety analysis set included all participants who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
Participants
  AEs | 11 | 16 | 16 | 12 | 55
  SAEs | 0 | 0 | 1 | 0 | 1

25. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included: systolic and diastolic blood pressure, heart rate, respiratory rate, percutaneous oxygen saturation, end-tidal carbon dioxide, core body temperature and body weight. Criteria for clinically significant vital signs abnormalities was based on Investigators decision.
Time Frame: Baseline up to 28 days after end of study drug dosing (Day 56)
Population: Safety analysis set included all participants who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
Participants | 0 | 0 | 0 | 0 | 0

26. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for abnormality: hemoglobin, hematocrit and red blood cell count <0.8*lower limit of normal(LLN); platelet <0.5*LLN; >1.75*upper limit of normal(ULN); white blood cell count <0.6*LLN; >1.5*ULN; lymphocytes, neutrophils and stab cells <0.8*LLN; >1.2*ULN; eosinophils, basophils and monocytes >1.2*ULN; total bilirubin >1.5*ULN; aspartate aminotransferase, alanine aminotransferase and gamma guanosine triphosphate and alkaline phosphatase >3*ULN; total protein and albumin <0.8*LLN; >1.2*ULN; glucose <0.6*LLN; >1.5*ULN; blood urea nitrogen and creatinine >1.3*ULN; uric acid >1.2*ULN; sodium <0.95*LLN; >1.05*ULN, potassium, calcium and magnesium <0.9*LLN; >1.1*ULN; phosphate <0.8*LLN; >1.2*ULN.
Time Frame: Baseline up to 28 days after end of study drug dosing (Day 56)
Population: Safety analysis set included all participants who received at least one dose of the investigational product. Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 18 | 12 | 62
Participants | 13 | 18 | 15 | 11 | 57

27. Other Pre Specified Outcome: Total Input/Output Fluid Volume
Description: Total input fluid volume was defined as the quantity of total fluids administered and total output fluid volume was defined as the quantity of total fluids excreted or lost during the specified evaluation period.
Time Frame: Baseline up to 28 days after end of study drug dosing (Day 56)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 18 | 12 | 63
milliliters (mL)
  Input Volume | 779.39 (342.617) | 799.18 (356.254) | 1023.60 (337.825) | 1415.96 (822.212) | 979.24 (520.514)
  Output Volume | 975.06 (436.904) | 801.53 (353.379) | 1041.80 (356.375) | 1313.58 (625.474) | 1009.58 (461.471)

28. Other Pre Specified Outcome: Incidence of Potential Withdrawal Symptoms
Description: The potential withdrawal symptoms were defined as AEs that occurred or worsened after end of administration of dexmedetomidine. It included bradycardia, abdominal discomfort, abdominal pain, dry mouth, nausea, vomiting, injection site pain, pyrexia, body temperature increased, electrocardiogram QT prolonged, neuralgia, agitation, atelectasis, oropharyngeal pain and hypotension. Incidence of potential withdrawal symptoms was reported in terms of number of participants who had any of the mentioned withdrawal symptoms.
Time Frame: Baseline up to 28 days after end of study drug dosing (Day 56)
Population: Safety analysis set included all participants who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
Participants
  Bradycardia | 0 | 4 | 0 | 0 | 4
  Abdominal discomfort | 0 | 0 | 1 | 0 | 1
  Abdominal pain | 0 | 0 | 0 | 1 | 1
  Dry mouth | 0 | 0 | 1 | 0 | 1
  Nausea | 0 | 0 | 2 | 3 | 5
  Vomiting | 1 | 1 | 1 | 4 | 7
  Injection site pain | 0 | 0 | 0 | 1 | 1
  Pyrexia | 1 | 0 | 0 | 0 | 1
  Body temperature increased | 1 | 0 | 0 | 0 | 1
  Electrocardiogram QT prolonged | 0 | 0 | 1 | 0 | 1
  Neuralgia | 0 | 0 | 0 | 1 | 1
  Agitation | 1 | 1 | 1 | 0 | 3
  Atelectasis | 1 | 1 | 0 | 0 | 2
  Oropharyngeal pain | 0 | 0 | 0 | 1 | 1
  Hypotension | 0 | 1 | 1 | 1 | 3

29. Other Pre Specified Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for clinically significant electrocardiogram abnormalities was based on Investigators decision.
Time Frame: Baseline up to 28 days after end of study drug dosing (Day 56)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
Number analyzed (Participants) | 14 | 18 | 19 | 12 | 63
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after end of study drug dosing (Day 56)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Dexmedetomidine: >=45 Weeks CGA to <12 Months | Dexmedetomidine: >=12 Months to <24 Months | Dexmedetomidine: >=2 Years to <6 Years | Dexmedetomidine: >=6 Years to <17 Years | Dexmedetomidine: All Participants
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18 | 0/19 | 0/12 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18 | 1/19 | 0/12 | 1/63
Other Adverse Events (participants affected / at risk) | 11/14 | 16/18 | 16/19 | 12/12 | 55/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine: >=45 Weeks CGA to <12 Months (N=14) | Dexmedetomidine: >=12 Months to <24 Months (N=18) | Dexmedetomidine: >=2 Years to <6 Years (N=19) | Dexmedetomidine: >=6 Years to <17 Years (N=12) | Dexmedetomidine: All Participants (N=63)
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine: >=45 Weeks CGA to <12 Months (N=14) | Dexmedetomidine: >=12 Months to <24 Months (N=18) | Dexmedetomidine: >=2 Years to <6 Years (N=19) | Dexmedetomidine: >=6 Years to <17 Years (N=12) | Dexmedetomidine: All Participants (N=63)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 6 | 7 | 5 | 2 | 20
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 5 | 9
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 2 | 1 | 2 | 6
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 5 | 7
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Body temperature increased (Investigations) | 1 | 2 | 0 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 4 | 2 | 1 | 0 | 7
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 3 | 5 | 17
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 3 | 8 | 11 | 9 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT02757625/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT02757625/SAP_001.pdf